CLINICAL TRIAL: NCT06680115
Title: Neoadjuvant and Adjuvant Sintilimab Combined with Chemoradiotherapy Versus Chemoradiotherapy Alone in Stage TanyN3M0 Nasopharyngeal Carcinoma: a Multicenter, Open-label, Randomized Phase II Clinical Trial
Brief Title: Neoadjuvant and Adjuvant Sintilimab Combined with Chemoradiotherapy Versus Chemoradiotherapy Alone in Stage TanyN3M0 Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-K395-01
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sintilimab (Experimental)
  Interventions: Drug: Sintilimab
- Control (No Intervention)

INTERVENTIONS:
Drug: Sintilimab — Induction chemotherapy stage: Sintilimab combined with GP regimen chemotherapy; Adjuvant chemotherapy stage: Sintilimab combined with Capecitabine
  Arms: Sintilimab

SUMMARY:
To evaluate the efficacy and safety of neoadjuvant and adjuvant Sintilimab combined with chemoradiotherapy versus chemoradiotherapy alone in stage TanyN3M0 nasopharyngeal carcinoma. The primary endpoint was 2-year failure-free survival (FFS). Secondary endpoints included 2-year overall survival (OS), distant failure-free survival (DFFS), locoregional failure-free survival (LRFFS), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma;
2. Age≥18 years;
3. Staging TanyN3M0 (AJCC/UICC 9th edition) ;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
5. White blood cell≥3.5×10^9/L,Neutrophils≥1.5×10^9/L, hemoglobin≥ 90 g/L, platelet (PLT)≥ 100x10^9/ L ;
6. Transaminases≤2.5 times the upper limit of normal, total bilirubin <1.5 times the upper limit of normal;
7. Creatinine clearance ≥60 ml/min;
8. Signed informed consent form.

Exclusion Criteria:

1. HBsAg positive and HBV DNA >1×103 copy/ml;
2. Patients with positive HCV antibody test results;
3. Active, known, or suspected autoimmune disease. Participants with type 1 diabetes, hypothyroidism requiring hormone replacement therapy, and skin conditions that do not require systemic treatment, such as vitiligo, psoriasis, or hair loss, may be enrolled;
4. History of interstitial lung disease;
5. Received systemic sex hormone or other immunosuppressive therapy with equivalent dose > 10mg prednisone/day within 28 days before signing the informed consent. Participants with a systemic sex hormone dose ≤10mg prednisone/day or inhaled/topical corticosteroids were enrolled;
6. Have received or will receive live vaccine within 30 days before signing the informed consent;
7. Pregnant or lactating women (pregnancy tests should be considered for sexually active, fertile women);
8. Had other malignancies within 5 years, except carcinoma in situ, adequately treated non-melanoma skin cancer, and papillary thyroid cancer;
9. The subject is known to have a prior allergy to macromolecular protein preparations, or any of the components of sindillizumab;
10. Human immunodeficiency virus (HIV) infection;
11. Other conditions, as determined by the investigator, that may affect subjects' safety or compliance with the study include symptomatic heart failure, unstable angina pectoris, myocardial infarction, active infection requiring systemic treatment, mental illness, or family and social factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
Distant failure-free survival | 2 years
Locoregional failure-free survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China